CLINICAL TRIAL: NCT00555607
Title: Longitudinal Assessment of Clinical Course and BIOmarkers in Severe Chronic AIRway Disease
Acronym: BIOAIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Athens (Other); University Hospital of Crete (Other); Università degli Studi di Ferrara (Other); University Ghent (Other); Pulmonary Research Institute Grosshansdorf (Unknown); Leiden University Medical Center (Other); Imperial College London (Other); Université Montpellier (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); University of Southampton (Other); Jagiellonian University (Other)
Responsible Party: Principal Investigator, Sven-Erik Dahlén, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIOAIR; QLG1-CT-2000-01185 (Other Grant/Funding Number: EU Fifth Framework Programe); FOOD-CT-2004-506378 (Other Grant/Funding Number: EU Sixth Framework Programme)
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Asthma; COPD
Keywords: asthma; COPD; severe; controlled; mild; biomarker; exacerbation
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lymphoma, Follicular | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- steroid (Active Comparator): Group receiving oral prednisolone (0.5 mg/kg bodyweight per day) during 14 days.
  Interventions: Drug: prednisolone
- placebo (Placebo Comparator): Group receiving placebo tablets during 14 days, followed by an open prednisolone treatment (0.5 mg/kg bodyweight per day) during a following 14 days.
  Interventions: Drug: prednisolone

INTERVENTIONS:
Drug: prednisolone — Prednisolone oral tablets (10 mg active ingredient per tablet) once a day at a dose of 0.5mg/kg bodyweight, during 14 days.

SUMMARY:
The aim of the project is to study pathogenetic mechanisms in severe asthma and compare those mechanisms in chronic obstructive pulmonary disease (COPD) in order to test the hypothesis that severe asthma and COPD develop into similar chronic degenerative changes.

DETAILED DESCRIPTION:
The BIOAIR project focuses on the sub-group of asthma patients that suffer from severe or difficult-to-control asthma, and who have frequent asthma exacerbations ('attacks'). This sub-group of asthma patients consists of around 10% of all asthma patients, but accounts for more than half of the total community costs for asthma. It is as yet unknown why these patients are so much more severely ill compared to the majority of asthma patients that have controlled disease. No adequate treatment has yet been established. The BIOAIR study was initiated in order to find out more about the mechanisms underlying severe asthma. Since some of the changes that occur in severe asthma are similar to patients with chronic obstructive lung disease (COPD), a group of COPD patients was included and will be studied as well. A group with controlled mild-to-moderate asthma was included for comparative reasons.

ELIGIBILITY:
Inclusion Criteria:

For all patients:

1. The patient understands the study procedures and agrees to participate by signing the consent form.
2. The patient is male or female, at least 18 years of age but no more than 80 years of age at the entry into the study (screening visit).

For patients with asthma (groups 1 and 2)

1. The patient has a history of intermittent or persistent symptoms of wheezing, breathlessness, chest tightness and cough. The diagnosis of asthma must have been confirmed by a specialist in pulmonary medicine.
2. The patient fulfils one or several of the following criteria for reversible airway obstruction, as documented during the last 5 years before the study or at screening visit:

   1. An increase in FEV1 more than 9% of predicted (or improvement by 200 mL) after administration of 4 puffs of 100 microg salbutamol dose-aerosol inhaler via a spacer, or after additional inhalation of four puffs of 20 microg ipratropium bromide (Atrovent) administered through a large volume spacer.
   2. A mean diurnal variation in Peak Expiratory Flow (PEF) of more than 15% on more than 4 days/week for at least 2 weeks, as calculated by the following equation:

      (highest PEF-lowest PEF)/mean PEF
   3. An increase in FEV1 of at least 400 mL after a course of prednisolone 0.5mg/kg/day for 14 days.
   4. In patients with a FEV1 more than 70% predicted, demonstrated bronchial hyperresponsiveness to histamine, methacholine, isocapnic hyperventilation, exercise or other indirect challenges (according to established local methods).
3. The patient is a non-smoker or has a total smoking history of less than 5 pack years. In the case the patient is smoking, it must be less than 10 cigarettes a day and the asthma must have started before smoking.

Specific for patients with mild to moderate asthma (group 1)

1. The patient has stable disease with minimal symptoms, no exacerbations or hospitalisations during the last year.
2. The patient uses inhaled steroids regularly, but not more than 800 microg/day budesonide or beclomethasone, or up to 500 microg/day fluticasone.
3. The patient uses prescribed short-acting beta agonists as needed.
4. The patient does not require treatment with long-acting beta-agonists.

Specific for patients with severe asthma (group 2)

1. The patient has been under specialist treatment for at least one year.
2. The patient requires continuous treatment with high doses of inhaled steroids. If the patient does not take oral steroids, the inhaled dose of steroids must be more than 1600 microg/day budesonide or beclomethasone, or more than 800 microg/day fluticasone or equivalent. In case the patient does take oral steroids, the inhaled dose of steroids must be more than 800 microg/day budesonide or beclomethasone, or more than 400 microg/day fluticasone or equivalent.
3. The patient requires continuous treatment with long acting inhaled beta-agonists or oral theophylline, as documented for at least one year.
4. The patient experienced at least one asthma exacerbation during the previous year.

Specific for patients with COPD (group 3)

1. The diagnosis of COPD must have been made by a specialist in pulmonary medicine. The patient may or may not have chronic symptoms (cough, sputum production, dyspnoea).
2. The patient has a FEV1/Forced Vital Capacity (FVC) ratio of less than 70%.
3. The patient's post bronchodilator FEV1 value is more than 30% but less than 80% of predicted.
4. The patient has a smoking history of more than 15 pack years, either as current or ex-smoker.
5. The patient displays a negative reversibility test to inhaled bronchodilators as defined by an increase in FEV1 of less than 9% of predicted (or an improvement by less than 200 mL) after administration of 4 puffs of 100 microg salbutamol dose-aerosol inhaler via a spacer, and four puffs of 20 microg ipratropium bromide (Atrovent) administered through a large volume spacer.
6. The patient has no history of asthma.
7. The patient has no current allergy, as shown by a negative skin-prick test.
8. The patient has used inhaled steroids in the range 800-1600 microg/day (budesonide or equivalent) for at least 3 months prior to the study.

Exclusion Criteria:

General exclusions

1. The patient is pregnant.
2. The patient has a recent history of incapacitating psychotic disorders.
3. The patient is a current or recent past abuser of alcohol or illicit drugs.
4. The patient has a history of malignancy, is known to be positive for HIV, or other states that are considered to interfere with study conduct or scientific interpretations.
5. The patient cannot read or comprehend written material, or is in the opinion of the investigator, for other reasons unlikely to understand and follow the study procedures.
6. The patient is mentally or legally incapacitated preventing informed consent from being obtained.

Exclusions because of pulmonary disorders

1. The patient is unable to perform acceptable spirometry, peak flow measurements and/or complete diary cards in a satisfactory way during the period between visit 1 and visit 3B (optimisation period and prednisolone/placebo trial). If the patient is unable to use the electronic Peak Flow meters/Diary cards, it is acceptable to use an ordinary mechanical meter (e.g. Mini-Wright) together with a paper version of the diary card. Patients that are unable to use the mechanical meter and paper diary card during the period between visit 1 and 3B cannot enter the follow-up year.
2. The patient has, in addition to asthma or COPD, any other pulmonary disorder that according to the investigator would interfere with the study procedures or scientific evaluation (e.g. tuberculosis).
3. The patient suffers from chronic hypercapnic respiratory failure as indicated by an elevated pCO2 (>47 mm Hg or 6,25 kPa). In case of doubt this should be confirmed with pulse oximetry or blood gas sampling.

Exclusions because of medications

1. The patient has received immunosuppressants other than corticosteroids (i.e., methotrexate, gold, troleandomycin, cyclosporin or any other experimental anti-inflammatory drug) within three months of study entry.
2. The patient is currently undergoing immunotherapy.
3. The patient receives chronic oxygen therapy.

Specific exclusion criterion for patients with asthma (groups 1 & 2)

1. The patient has smoked more than five (5) pack years.

Specific exclusion criterion for patients with mild asthma (group 1) 1. The patient requires treatment with long-acting beta-agonists.

Specific exclusion criteria for patients with severe asthma (group 2)

1. The patient is not treated with high doses of inhaled steroids (see above).
2. The patient has not had an exacerbation of asthma during the last year.
3. The patient does not require treatment with long-acting beta-agonists or theophylline as documented during one year.

Specific exclusion criterion for patients with COPD (group 3)

1. The patient has a history of asthma confirmed by a specialist in pulmonary medicine.

Specific exclusion criteria for bronchoscopy (all groups)

1. The patient has had a severe exacerbation of asthma requiring high doses of oral steroids during the last three (3) months.
2. The patient has had a severe exacerbation of COPD requiring intensive outpatient treatment or hospitalisation during the last three (3) months.
3. The patient has had three or more severe exacerbations of asthma or COPD during the last year.
4. The patient displays more than 10% fall in FEV1 at 2 minutes after inhalation of 0.9% saline (during induction of sputum at visit 2).
5. The patient has shown signs of uncontrolled disease during the last three days, e.g. the patient has required more than four puffs/day of rescue medication above baseline use during the last three days. (In the case criteria 1-4 are not met, such patients may be rescheduled for bronchoscopy in two weeks time. The start of the oral prednisolone intervention will then be postponed by the number of days passing before the bronchoscopy).
6. If a patient who otherwise has qualified for bronchoscopy has received more than 6 mg per kg BW of lidocaine during the preparation for the procedure, the bronchoscopy must be terminated and cannot be continued the same day.
7. Patients who have experienced severe bronchoconstriction or other adverse reactions at previous attempts to perform bronchoscopy.
8. The patient has a post-bronchodilator FEV1 < 40% predicted.
9. Do not start or proceed bronchoscopy if:

   * Transcutaneous oxygen saturation by pulse-oximeter < 90% (despite giving oxygen by nasal cannula when saturation is < 94%)
   * Heart frequency > 130
   * Heart rhythm disturbances.

Specific exclusion criteria for induced sputum (all groups)

1. A post-bronchodilator (after administration of 4 puffs of 100 microg salbutamol dose-aerosol inhaler via a spacer) FEV1 percent of predicted being less than 60%, or in absolute values less than 1.0 L.
2. A peak flow variability of more than 30% during the previous four days.
3. Patients who display more than a 15% fall in FEV1 at 2 minutes after inhalation of saline (0.9% NaCl) during induction of sputum..
4. Patients who have experienced severe bronchoconstriction or other adverse reactions at previous attempts to induce sputum.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2002-03; Primary Completion 2005-04 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of exacerbations | one year

SECONDARY OUTCOMES:
Steroid responsiveness | 2 weeks
Lung function (Peak Expiratory Flow) | one year
Biomarkers | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Dahlén, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Kupczyk M, Haque S, Middelveld RJ, Dahlen B, Dahlen SE; BIOAIR Investigators. Phenotypic predictors of response to oral glucocorticosteroids in severe asthma. Respir Med. 2013 Oct;107(10):1521-30. doi: 10.1016/j.rmed.2013.07.014. Epub 2013 Aug 27. PMID 23993706
- See also: Related Info — http://www.ist-world.org/ProjectDetails.aspx?ProjectId=b3da9185132d491487bd61f995ac89e8&SourceDatabaseID=9cd97ac2e51045e39c2ad6b86dce1ac2